CLINICAL TRIAL: NCT07289464
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of RSS0343 Following Multiple Oral Doses in Healthy Subjects, as Well as Its Effects on the QT/QTc Interval
Brief Title: A Clinical Study of RSS0343 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSS0343-102
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSS0343 Tablets Group (Experimental)
  Interventions: Drug: RSS0343 Tablets
- RSS0343 Tablets Placebo Group (Placebo Comparator)
  Interventions: Drug: RSS0343 Tablets Placebo

INTERVENTIONS:
Drug: RSS0343 Tablets — RSS0343 tablets, oral.
  Arms: RSS0343 Tablets Group
Drug: RSS0343 Tablets Placebo — RSS0343 tablets placebo, oral.
  Arms: RSS0343 Tablets Placebo Group

SUMMARY:
This is a phase I study to evaluate the safety, tolerability and pharmacokinetics of RSS0343 following multiple oral doses in healthy subjects, as well as its effects on the QT/QTc interval.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provided written informed consent after being fully informed of the trial's purpose, significance, and protocol requirements.
2. Healthy individuals aged 18 to 55 years, inclusive. Males and females
3. Body weight ≥ 50 kg for males and ≥ 45 kg for females. Body mass index (BMI) = weight (kg)/height 2 (m²). BMI between 19 and 28 kg/m², inclusive.
4. Fertile male and female subjects and their partners must agree to use highly effective contraception as stipulated in the protocol, from screening until 6 months (for females) or 3 months (for males) after the last dose. Additionally, fertile female subjects must have a negative serum pregnancy test at screening and prior to the first dose (baseline) and must not be lactating.

Exclusion Criteria:

1. Subjects who smoked more than 5 cigarettes (or equivalent nicotine products) daily within 3 months prior to screening or intended to use tobacco products during the trial.
2. Subjects with frequent alcohol consumption (>15 g/day for females or >25 g/day for males [5g of alcohol is equivalent to 150 mL of beer, 50 mL of wine or approximately 17 mL of low-alcohol liquor], on more than 2 occasions per week) within 6 months prior to screening, or were unable to abstain during the trial, or who tested positive on the alcohol breath test at baseline.
3. Subjects with a history of, or current, drug abuse, or drug dependence (during consultation), or with a positive urine drug screening result.
4. Subjects who had donated blood or experienced a total blood loss of ≥200 mL within 1 month, or ≥400 mL within 3 months prior to dosing, or who had received a blood transfusion within 8 weeks prior to dosing.
5. Subjects with dysphagia; or a history of needle or blood phobia, poor venous access, or inability to tolerate venipuncture.
6. Subjects deemed by the investigators to be unsuitable for the trial for any other reason.
7. Subjects with any clinically significant abnormalities, as determined by the investigator, in physical examination, vital signs, laboratory tests (including hematology, urinalysis, blood biochemistry, coagulation), chest imaging, abdominal ultrasonography, or electrocardiogram.
8. Subjects who tested positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or HIV antibody.
9. Subjects with a known or suspected allergy to the investigational drug or its excipients, or a history of severe allergic reactions (e.g., to drugs, food, toxins).
10. Subjects with any active autoimmune disease or immunodeficiency at screening.
11. Subjects with any history of severe clinical disease, or any condition that, in the investigator's judgment, could compromise trial outcomes, affect drug absorption, distribution, metabolism, or excretion (pharmacokinetics), or pose an undue risk to the subject. This includes, but is not limited to, significant disorders of the circulatory, endocrine, nervous, digestive, urinary, hematological, immune, psychiatric, or metabolic systems.
12. Subjects who had undergone any surgery within 3 months prior to screening, had not fully recovered as determined by the investigator, or planned to undergo surgery during the trial or within 1 month after its completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of any adverse events (AEs). | Evaluation was performed up to Day 28.
  Safety and tolerability.

SECONDARY OUTCOMES:
Maximum observed plasma concentration of RSS0343 at Day 1 (Cmax). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Maximum observed plasma concentration of RSS0343 at steady state (Cmax,ss). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Time to Cmax (Tmax). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Time to Cmax,ss (Tmax,ss). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Area under the concentration-time curve during a dosing interval (AUC0-tau). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Area under the concentration-time curve from 0 to the last measurable time point after RSS0343 administration (AUC0-t). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Area under the concentration-time curve from time 0 to infinity after RSS0343 administration (AUC0-inf). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Terminal elimination half-life of RSS0343 (t1/2). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Apparent clearance of RSS0343 during multiple dosing with a dosing interval of time tau (CLss/F). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Apparent volume of distribution during terminal elimination phase of RSS0343 at steady state (Vss/F). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Cumulative amount of drug excreted in urine (Ae,urine). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Cumulative percentage of dose recovered in urine (Fe,urine). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Renal clearance of RSS0343 (CLr). | Evaluation was performed up to Day 28.
  Pharmacokinetics (PK) indicator.
Changes in the QTc interval corrected by the Fridericia method relative to baseline (ΔQTcF) (where applicable). | Evaluation was performed up to Day 28.
  To evaluate the effects of RSS0343 on the QT/QTc interval in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided